CLINICAL TRIAL: NCT02524860
Title: Targeted Prostate Biopsy Using a Novel MRI-Ultrasound Fusion Device in Patients With an Elevated PSA and a Positive Multiparametric MRI
Brief Title: Targeted Prostate Biopsy Using a Novel MRI-Ultrasound Fusion Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Focal Healthcare Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150330, version 2.0
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Biopsy; Focal Healthcare; Fusion Targeted Biopsy; High Risk Cancer; Imaging; Diagnostic; Ultrasound; Multiparametric Magnetic Resonance Imaging (MP-MRI); MRI-Ultrasound Fusion; Focal-Fusion Bx
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI-ultrasound fusion device (Experimental): Using the Focal-Fusion Bx device, the urologist will fuse ('coregister') the MRI to the TRUS imaging
  Interventions: Device: Focal-Fusion Bx

INTERVENTIONS:
Device: Focal-Fusion Bx — The Focal-Fusion Bx device uses hardware and software to overlay targets onto the live ultrasound image in real-time. This allows the urologist to take biopsy samples from tissue that looked suspicious on the patient's MRI.
  Other Names: MRI-ultrasound fusion device

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Focal-Fusion Bx at detecting clinically significant prostate cancer in a standard clinical environment.

DETAILED DESCRIPTION:
The objective of this study is to determine the effectiveness of the Focal-Fusion Bx device at finding clinically relevant prostate cancer.

A multiparametric MRI examination will be carried out prior to study enrollment. Probable cancerous regions (regions of interest, ROI) will be identified, and these ROIs will be used as targets during the biopsy.

Three prostate sampling methods will be conducted in the same session on all patients. These include:

i) Focal-Fusion Bx targeted biopsy ii) Cognitive fusion targeted biopsy and iii) Systematic (untargeted) biopsy. Trans-rectal ultrasound (TRUS) imaging will be conducted with BK Flex Focus Ultrasound system (Analogic Corporation, Peabody, MA).

Primary hypothesis: The technique used to acquire the biopsy samples will impact the proportion of clinically relevant cancers by improving the specificity of detecting clinically significant cancers. It is hypothesized that Focal-Fusion Bx biopsies will diagnose more high risk cancers and fewer low-risk cancers than non-targeted systematic biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subjects up to 80 years of age
* Candidates for fusion biopsy
* Elevated PSA levels
* MP-MRI with lesions having a Prostate Imaging Reporting and Data System (PI-RADS) score greater than or equal to 3 (determined by a trained radiologist)
* Subject is willing and able to read, understand and sign the Informed Consent Form document

Exclusion Criteria:

* Previous treatment for prostate cancer
* Any contraindication to a standard TRUS prostate biopsy procedure
* Refusal to sign the Informed Consent document

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of biopsy cores positive for clinically significant cancer. | 12 months

SECONDARY OUTCOMES:
Number of men diagnosed with clinically significant and clinically insignificant cancer. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Winston Barzell, MD, Principal Investigator — 21st Century Oncology, Inc.
Locations (1):
- Urology Treatment Center (division of 21st Century Oncology, Inc.), Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided